CLINICAL TRIAL: NCT05093075
Title: Therapeutic Plasma Exchange in Septic Shock: A Pilot Study
Acronym: PLEXSIS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Health Sciences Centre Foundation, Manitoba (Other); McMaster University (Other); University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS23165 (B2019:093)
Record Dates: First submitted 2021-07-19; First posted 2021-10-26 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Septic Shock
Keywords: Sepsis
MeSH Terms: conditions — Shock, Septic; Sepsis | interventions — Plasma Exchange

STUDY DESIGN:
Intervention Model Description: A web-based randomization system maintained at the Center for Healthcare Innovation (CHI) (Winnipeg, Manitoba) will be used to allocate treatment assignments. The randomization process will consist of a computer-generated random listing of the treatment allocations in variable permuted blocks of 2 and 4. Participants will be randomized to Treatment (5 Therapeutic Plasma Exchanges) or Standard of Care.
Who Masked: Investigator, Outcomes Assessor
Masking Description: All investigators and research staff will be blinded to the allocation schedules. The PLEXSIS pilot trial is designed as a prospective randomized open, blinded endpoint (PROBE) trial. This pragmatic design is necessary given impractical nature of blinding the TPE intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Arm (Experimental): Participants randomized to the Treatment Arm will received 1.0 plasma exchanges daily until discontinuation of vasopressors, death or to a maximum of 5 daily treatments. Solvent detergent plasma (SDP) or frozen plasma (FP) depending on availability will be used as the replacement fluid.
  Interventions: Other: Therapeutic Plasma Exchange
- Standard of Care Arm (No Intervention): Participants randomized to the Control Arm will receive standard of care for the treatment of septic shock in accordance with local practice and informed by national and international guidelines.

INTERVENTIONS:
Other: Therapeutic Plasma Exchange — TPE procedures will be performed using a Spectra Optia ® apheresis machine (Terumo BCT, Lakewood, USA) according to usual-care procedures for apheresis. Venous access for the TPE procedures will be obtained through a double lumen dialysis catheter to provide adequate flow rates required for TPE. Regional citrate anticoagulation will be used for anticoagulation within the apheresis circuit. One to two grams of calcium chloride will be infused as per standard during TPE to prevent symptomatic hypocalcemia. Plasma volume will be calculated as per a standard formula whereby estimated plasma volume (in liters) = 0.07 x weight (kg) x (1 - hematocrit). In patients on dialysis, dialysis will be interrupted for the duration of the procedure. Antibiotics will be given after TPE to avoid clearance of the antibiotics. On the first day of TPE, a repeat dose of antibiotics will be administered after completion of TPE. Nurse clinicians trained in TPE will perform the TPE procedures.
  Arms: Treatment Arm

SUMMARY:
The investigators propose to conduct a multi-center randomized pilot feasibility trial comparing therapeutic plasma exchange to standard of care in patients diagnosed with septic shock.

DETAILED DESCRIPTION:
The intervention arm consists of an exchange of one volume of plasma equivalent to the patient's total calculated blood volume (1.0 plasma volume exchange) performed daily until discontinuation of vasopressors, death or up to a maximum of 5 daily treatments. Solvent detergent plasma or frozen plasma (FP) depending on availability will be used as the replacement fluid. The control group will receive standard of care for the treatment of septic shock in accordance with local practice and informed by national and international guidelines.

The management of septic shock, including but not limited to, antibiotic therapy, infection source control, therapy, fluid therapy, mechanical ventilation, and nutrition, will be at the discretion of the treating medical team, and will be recorded and reported.

The investigators will monitor for development of coagulopathy by measure the INR and fibrinogen levels daily. These are expected to normalize with the use of plasma as replacement fluid. The investigators will monitor for adverse reactions related to central venous access devices (insertion related complications, infection, thrombosis) and/or TPE (including reaction to plasma, allergic reactions and hypotension). Venous access devices will be inserted by trained, experienced personnel using real-time ultrasound guidance. These data are routinely collected by apheresis programs across Canada as part of a data collection and reporting relationship with CAG.

To further our understanding of the biologic impact of TPE in sepsis, plasma and whole blood samples will be collected at randomization (day 1), Pre-3rd TPE or Day 3 if in SOC group, pre-5th TPE or Day if SOC group, and 48 hours after completion of TPE or Day 7 if SOC group to evaluate markers of coagulation (ADAMTS-13 levels, DNase levels, histones).

ELIGIBILITY:
Eligible patients must be admitted to an ICU and must meet all of the following inclusion criteria:

1. ≥ 16 years of age
2. Refractory hypotension documented within 48 hours prior to enrollment requiring the institution and ongoing use of vasopressor agents (phenylephrine, norepinephrine, vasopressin, epinephrine, midodrine or dopamine >5 mcg/kg/min) at enrollment. Refractory hypotension is defined as a systolic blood pressure (SBP) less than 90 mmHg, or SBP less than 30 mmHg below baseline, or a mean arterial blood pressure less than 65 mmHg, despite adequate fluid resuscitation
3. Capacity to initiate plasma exchange with 48 hours of vasopressor initiation.
4. At least 1 other new organ dysfunction (in addition to refractory hypotension), defined by the following at the time of enrollment:

   1. Creatinine ≥1.5x the known baseline creatinine within 7 days, or ≥ 26.5 µmol/l increase in 48 hours,
   2. Need for invasive mechanical ventilation or a P/F ratio <250
   3. Platelets <100 x109/L, or a drop of 50 x109/L in the 3 days prior to enrollment
   4. Arterial pH < 7.30 or base deficit > 5 mmol/L in association with a lactate >/= to 3.0 mmol/L

45. Known or suspected infection

2.4.3 Exclusion criteria

We will exclude patients who have any one of the following criteria at the time of enrollment:

1. Consent declined (refusal from patient, SDM, or physician)
2. Clinically apparent alternate causes for shock (cardiogenic, hemorrhagic, obstructive, neurogenic or anaphylactic)
3. Terminal illness with a life expectancy of less than 3 months
4. Are pregnant

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Assess the feasibility of a large, multicenter trial of TPE in patients with septic shock | 18 months for enrollment
  Assessing the feasibility of a large, multicenter trial of TPE in patients with septic shock will be the primary outcome. The primary measure of feasibility will be the ability to enroll an average of 2 patients per site per month.

SECONDARY OUTCOMES:
Assess the rate of enrollment and adherence to the protocol of those enrolled | 18 months
  The investigators will consider the consent rate to be adequate if 70% of SDM or patients when approached for consent are enrolled, an acceptable rate of protocol adherence to be 90% of all study participants; and the time from randomization to study treatment initiation to be satisfactory if this interval is less than 24 hours.
Number of participants that develop adverse reactions to TPE | Up to 8 days
  The following will be recorded: a) major respiratory compromise; b) thrombotic events; c) major bleeding; d) anaphylaxis; e) central venous access insertion complications.
Further understand the biological impact of TPE in sepsis | up to 8 days
  To further our understanding of the biologic impact of TPE in sepsis, sites will collect plasma and whole blood samples at randomization (day 1), pre-3rd TPE or day 3 if in SOC group, pre-5th TPE or day 5 if SOC group, and 48 hours after completion of last TPE or day 7 if SOC group to evaluate markers of coagulation (ADAMTS-13 levels, DNase levels, histones). Sites will collect whole blood samples on all randomized patients and profile DNA methylation on a random subset of 40 patients to determine changes in circulating immune cell remodeling.

OTHER OUTCOMES:
Mortality | up to day 60
  The pilot trial is not designed to detect differences in clinical outcomes. However, vital status will be accessed.
Organ failure | Up to day 21
  The pilot trial is not designed to detect differences in clinical outcomes. However, the investigators will measure and describe organ-support free-days to day 21, and change in SOFA score (multiple organ dysfunction score).
Organ failure | Up to day 8
  The pilot trial is not designed to detect differences in clinical outcomes. However, the investigators will measure change in SOFA score (multiple organ dysfunction score).

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Zarychanski, MD, MSc, Principal Investigator — University of Manitoba; Emily Rimmer, MD, MSc, Principal Investigator — University of Manitoba
Locations (11):
- Canada (11):
  - Foothills Medical Centre, Calgary, Alberta
  - Southern Health Campus, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - University of Manitoba, Winnipeg, Manitoba
  - Hamilton Health Sciences - Juravinski, Hamilton, Ontario
  - St. Joseph's Hospital, Hamilton, Ontario
  - Queen's University at Kingston, Kingston, Ontario
  - Ottawa Hospital, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Centre Hospitalier de L'Université de Montréal (Chum),, Montreal, Quebec
  - Universite Laval, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No
The investigators do not plan to make individual participant data available to other researchers.

REFERENCES:
- [Background] Schwartz J, Padmanabhan A, Aqui N, Balogun RA, Connelly-Smith L, Delaney M, Dunbar NM, Witt V, Wu Y, Shaz BH. Guidelines on the Use of Therapeutic Apheresis in Clinical Practice-Evidence-Based Approach from the Writing Committee of the American Society for Apheresis: The Seventh Special Issue. J Clin Apher. 2016 Jun;31(3):149-62. doi: 10.1002/jca.21470. PMID 27322218
- [Background] Rimmer E, Houston BL, Kumar A, Abou-Setta AM, Friesen C, Marshall JC, Rock G, Turgeon AF, Cook DJ, Houston DS, Zarychanski R. The efficacy and safety of plasma exchange in patients with sepsis and septic shock: a systematic review and meta-analysis. Crit Care. 2014 Dec 20;18(6):699. doi: 10.1186/s13054-014-0699-2. PMID 25527094
- [Background] Busund R, Koukline V, Utrobin U, Nedashkovsky E. Plasmapheresis in severe sepsis and septic shock: a prospective, randomised, controlled trial. Intensive Care Med. 2002 Oct;28(10):1434-9. doi: 10.1007/s00134-002-1410-7. Epub 2002 Jul 23. PMID 12373468
- [Background] Davies R, O'Dea K, Gordon A. Immune therapy in sepsis: Are we ready to try again? J Intensive Care Soc. 2018 Nov;19(4):326-344. doi: 10.1177/1751143718765407. Epub 2018 Apr 4. PMID 30515242
- [Background] Dellinger RP, Levy MM, Carlet JM, Bion J, Parker MM, Jaeschke R, Reinhart K, Angus DC, Brun-Buisson C, Beale R, Calandra T, Dhainaut JF, Gerlach H, Harvey M, Marini JJ, Marshall J, Ranieri M, Ramsay G, Sevransky J, Thompson BT, Townsend S, Vender JS, Zimmerman JL, Vincent JL; International Surviving Sepsis Campaign Guidelines Committee; American Association of Critical-Care Nurses; American College of Chest Physicians; American College of Emergency Physicians; Canadian Critical Care Society; European Society of Clinical Microbiology and Infectious Diseases; European Society of Intensive Care Medicine; European Respiratory Society; International Sepsis Forum; Japanese Association for Acute Medicine; Japanese Society of Intensive Care Medicine; Society of Critical Care Medicine; Society of Hospital Medicine; Surgical Infection Society; World Federation of Societies of Intensive and Critical Care Medicine. Surviving Sepsis Campaign: international guidelines for management of severe sepsis and septic shock: 2008. Crit Care Med. 2008 Jan;36(1):296-327. doi: 10.1097/01.CCM.0000298158.12101.41. PMID 18158437
- [Background] Lega JC, Mismetti P, Cucherat M, Fassier T, Bertoletti L, Chapelle C, Laporte S. Impact of double-blind vs. open study design on the observed treatment effects of new oral anticoagulants in atrial fibrillation: a meta-analysis. J Thromb Haemost. 2013 Jul;11(7):1240-50. doi: 10.1111/jth.12294. PMID 23659614
- [Background] Binnie A, Walsh CJ, Hu P, Dwivedi DJ, Fox-Robichaud A, Liaw PC, Tsang JLY, Batt J, Carrasqueiro G, Gupta S, Marshall JC, Castelo-Branco P, Dos Santos CC; Epigenetic Profiling in Severe Sepsis (EPSIS) Study of the Canadian Critical Care Translational Biology Group (CCCTBG). Epigenetic Profiling in Severe Sepsis: A Pilot Study of DNA Methylation Profiles in Critical Illness. Crit Care Med. 2020 Feb;48(2):142-150. doi: 10.1097/CCM.0000000000004097. PMID 31939781